CLINICAL TRIAL: NCT05305170
Title: Plasmatic Levels of Epoxyeicosatrienoic and Dihydroxyeicosatrienoic Acids in Heart Failure
Brief Title: Eicosanoids in Human Heart Failure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Motol (Other)
Responsible Party: Principal Investigator, Petr Kala, MD, Petr Kala, MD, University Hospital, Motol
Other Study IDs: UHMotol
Record Dates: First submitted 2022-03-22; First posted 2022-03-31 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-03

CONDITIONS: Heart Failure
Keywords: heart failure; eicosanoids; reverse remodeling
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HF: Patients with heart failure.
  Interventions: Diagnostic Test: Levels of EETs, DHETs and HETEs
- Controls: Controls without heart failure.
  Interventions: Diagnostic Test: Levels of EETs, DHETs and HETEs

INTERVENTIONS:
Diagnostic Test: Levels of EETs, DHETs and HETEs — The plasmatic concentration of EETs, DHETs, and HETEs.

SUMMARY:
Our translational project aims to evaluate the role of eicosanoids in human HF.

DETAILED DESCRIPTION:
Heart failure (HF) is the leading cause of cardiovascular hospitalizations, and with its increasing prevalence, the healthcare systems face a heart failure pandemic. Translational research findings improve our knowledge of pathophysiology and uncover therapeutic targets in HF. Natriuretic peptides represent such examples as routinely used in diagnostics and therapeutics (neprilysin inhibitor). Despite modern pharmacotherapy, including angiotensin receptor-neprilysin inhibitor (ARNI) and sodium-glucose cotransporter-2 inhibitors (SGLT2i), the prognosis of patients, especially with advanced heart failure, remains poor. Furthermore, most medication is limited in the late stages of HF due to their hypotensive effects.

Basic research has been focused on the eicosanoids - metabolites of cytochrome P-450 (CYP)-dependent epoxygenase pathway of arachidonic acid (AA), especially epoxyeicosatrienoic acids (EETs). In the preclinical studies, it was shown that EETs importantly contribute to the regulation of cardiovascular and renal function and exert organ-protective actions. It was also proposed that intrarenal EETs operate as an endogenous compensatory system opposing increased renin-angiotensin system (RAS) activity. EETs are rapidly transformed by soluble epoxide hydrolase (sEH) to biologically inactive dihydroxyeicosatrienoic acids (DHETs). The role of eicosanoids in human HF, however, remains unclear.

Our translational project (Eicosanoids in Human Heart Failure) aims to evaluate the role of eicosanoids in human HF.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart failure patients from our tertiary cardiovascular center and controls from the central hospital laboratory.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasmatic levels of eicosanoids | at enrollment
  EET, DHET, 20-HETE

SECONDARY OUTCOMES:
Mortality | 2 years
  Overall mortality

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Motol, Prague, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Conrad N, Judge A, Tran J, Mohseni H, Hedgecott D, Crespillo AP, Allison M, Hemingway H, Cleland JG, McMurray JJV, Rahimi K. Temporal trends and patterns in heart failure incidence: a population-based study of 4 million individuals. Lancet. 2018 Feb 10;391(10120):572-580. doi: 10.1016/S0140-6736(17)32520-5. Epub 2017 Nov 21. PMID 29174292
- [Background] McDonagh TA, Metra M, Adamo M, Gardner RS, Baumbach A, Bohm M, Burri H, Butler J, Celutkiene J, Chioncel O, Cleland JGF, Coats AJS, Crespo-Leiro MG, Farmakis D, Gilard M, Heymans S, Hoes AW, Jaarsma T, Jankowska EA, Lainscak M, Lam CSP, Lyon AR, McMurray JJV, Mebazaa A, Mindham R, Muneretto C, Francesco Piepoli M, Price S, Rosano GMC, Ruschitzka F, Kathrine Skibelund A; ESC Scientific Document Group. 2021 ESC Guidelines for the diagnosis and treatment of acute and chronic heart failure. Eur Heart J. 2021 Sep 21;42(36):3599-3726. doi: 10.1093/eurheartj/ehab368. No abstract available. PMID 34447992
- [Background] Vaduganathan M, Claggett BL, Jhund PS, Cunningham JW, Pedro Ferreira J, Zannad F, Packer M, Fonarow GC, McMurray JJV, Solomon SD. Estimating lifetime benefits of comprehensive disease-modifying pharmacological therapies in patients with heart failure with reduced ejection fraction: a comparative analysis of three randomised controlled trials. Lancet. 2020 Jul 11;396(10244):121-128. doi: 10.1016/S0140-6736(20)30748-0. Epub 2020 May 21. PMID 32446323
- [Background] Imig JD, Cervenka L, Neckar J. Epoxylipids and soluble epoxide hydrolase in heart diseases. Biochem Pharmacol. 2022 Jan;195:114866. doi: 10.1016/j.bcp.2021.114866. Epub 2021 Dec 2. PMID 34863976
- [Background] Fan F, Roman RJ. Effect of Cytochrome P450 Metabolites of Arachidonic Acid in Nephrology. J Am Soc Nephrol. 2017 Oct;28(10):2845-2855. doi: 10.1681/ASN.2017030252. Epub 2017 Jul 12. PMID 28701518
- [Background] Jamieson KL, Endo T, Darwesh AM, Samokhvalov V, Seubert JM. Cytochrome P450-derived eicosanoids and heart function. Pharmacol Ther. 2017 Nov;179:47-83. doi: 10.1016/j.pharmthera.2017.05.005. Epub 2017 May 25. PMID 28551025
- [Background] Elmarakby AA. Reno-protective mechanisms of epoxyeicosatrienoic acids in cardiovascular disease. Am J Physiol Regul Integr Comp Physiol. 2012 Feb 1;302(3):R321-30. doi: 10.1152/ajpregu.00606.2011. Epub 2011 Nov 23. PMID 22116511
- [Background] Sporkova A, Reddy RN, Falck JR, Imig JD, Kopkan L, Sadowski J, Cervenka L. Interlobular Arteries From 2-Kidney, 1-Clip Goldblatt Hypertensive Rats' Exhibit-Impaired Vasodilator Response to Epoxyeicosatrienoic Acids. Am J Med Sci. 2016 May;351(5):513-9. doi: 10.1016/j.amjms.2016.02.030. Epub 2016 Feb 23. PMID 27140711
- [Background] Fleming I. The pharmacology of the cytochrome P450 epoxygenase/soluble epoxide hydrolase axis in the vasculature and cardiovascular disease. Pharmacol Rev. 2014 Oct;66(4):1106-40. doi: 10.1124/pr.113.007781. PMID 25244930
- [Background] Imig JD, Elmarakby A, Nithipatikom K, Wei S, Capdevila JH, Tuniki VR, Sangras B, Anjaiah S, Manthati VL, Sudarshan Reddy D, Falck JR. Development of epoxyeicosatrienoic acid analogs with in vivo anti-hypertensive actions. Front Physiol. 2010 Dec 3;1:157. doi: 10.3389/fphys.2010.00157. eCollection 2010. PMID 21423396
- [Background] Gawrys O, Huskova Z, Baranowska I, Walkowska A, Sadowski J, Kikerlova S, Vanourkova Z, Honetschlagerova Z, Skaroupkova P, Cervenka L, Falck JR, Imig JD, Kompanowska-Jezierska E. Combined treatment with epoxyeicosatrienoic acid analog and 20-hydroxyeicosatetraenoic acid antagonist provides substantial hypotensive effect in spontaneously hypertensive rats. J Hypertens. 2020 Sep;38(9):1802-1810. doi: 10.1097/HJH.0000000000002462. PMID 32384390
- [Background] Kala P, Miklovic M, Jichova S, Skaroupkova P, Vanourkova Z, Maxova H, Gawrys O, Kompanowska-Jezierska E, Sadowski J, Imig JD, Falck JR, Veselka J, Cervenka L, Aiglova R, Vicha M, Gloger V, Taborsky M. Effects of Epoxyeicosatrienoic Acid-Enhancing Therapy on the Course of Congestive Heart Failure in Angiotensin II-Dependent Rat Hypertension: From mRNA Analysis towards Functional In Vivo Evaluation. Biomedicines. 2021 Aug 20;9(8):1053. doi: 10.3390/biomedicines9081053. PMID 34440257